CLINICAL TRIAL: NCT02518945
Title: Dapagliflozin As Additional Treatment To Liraglutide And Insulin In Patients With Type 1 Diabetes. A Randomized Clinical Trial
Brief Title: Dapagliflozin As Additional Treatment To Liraglutide And Insulin In Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1969
Record Dates: First submitted 2015-07-31; First posted 2015-08-10 (Estimated); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Liraglutide; Dapagliflozin; Triple Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin; Insulin; Insulin Glargine; Insulin Detemir; Insulin Lispro; Insulin Aspart; insulin glulisine; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 12 weeks of treatment with Insulin, Liraglutide and "Dapagliflozin Placebo"
  Interventions: Drug: Insulin; Drug: Liraglutide; Drug: Dapagliflozin placebo
- Active drugs (Active Comparator): 12 weeks of treatment with Insulin, Liraglutide and "Active Dapagliflozin Drug"
  Interventions: Drug: Dapagliflozin; Drug: Insulin; Drug: Liraglutide

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin or Farxiga is a SGLT-2 inhibitor
  Other Names: Farxiga
  Arms: Active drugs
Drug: Insulin
  Other Names: Lantus, Levemir, Toujjeo, Humalog , Novolog, Apidra
Drug: Liraglutide — Victoza(Liraglutide) is a GLP-1 agent.
  Other Names: Victoza
Drug: Dapagliflozin placebo — Dapagliflozin placebo looking similar to active drug Dapagliflozin in external appearance but not containing active ingredient dapagliflozin
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a single center, prospective, randomized, double blinded placebo controlled study conducted I patients with type 1 diabetes.The aim of this study is to examine the additive effects of GLP-1 agonist and SGLT2 inhibitor in patients with type 1 diabetes in terms of possible improved glycemic control, reduced glycemic variability, reduced insulin dosages, additional effects of weight loss and blood pressure reduction.

DETAILED DESCRIPTION:
This investigation will be single center, prospective, randomized, double blinded placebo controlled study conducted in type 1 diabetics. The study will be conducted at Diabetes - Endocrinology Center of WNY, affiliated to the State University of New York at Buffalo.

Visit 1: Screening Day (day -21):- Each patient will have completed the following procedures prior to participating in the study.

1. Medical History;
2. Physical Exam;
3. Informed consent.
4. Baseline lab draws to measure CBC, comprehensive metabolic panel, Hba1c, Fructosamine and lipid profile. All labs will be drawn in the fasting state in the morning before 10am.

Visit 2: Randomization Visit (day -14): After the screening visit, subjects who meet the inclusion and exclusion criteria will participate in the study period. Randomization will be done by a ratio of 2:1(drug: placebo) using Microsoft Excel randomization function. Liraglutide will be obtained from Novo Nordisk pharmaceuticals. Dapagliflozin/placebo will be obtained from Astra Zeneca pharmaceuticals. All subjects will be instructed by the study staff in the dosing and administration of the study medication. Subjects will be seen by a registered dietitian who will review their carbohydrate counting and make an assessment of their carbohydrate intake. A CGM sensor will be inserted and the patient will be asked to keep it for 2 weeks. Detailed instruction on changing the sensor weekly will be provided and insulin titration will be done to control blood sugar between 70-180 mg/dl. A urine container to collect urine for 24 hours to measure 24-hour urinary glucose will be provided (urine to be collected one day before the next visit).

All subjects will be advised to monitor their capillary blood glucose by finger stick before each meal and at bedtime and to wear their CGM constantly for the first two weeks and the last two weeks of the study The subjects will be asked to keep a diary of their food intake to measure their carbohydrate intake. For the entire duration of the study, the patients will maintain a diary to record any hypoglycemia and other untoward side effects like nausea, changes in appetite and other experiences. Patients will be instructed to call the Diabetes Center or an endocrinology fellow directly in case of any problem or untoward side effects. They will be specifically asked to call if they have hypoglycemia (blood sugar <70 mg/dl) or hyperglycemia (blood sugar >250 mg/dl) on more than one occasion.

Visit 3 Study Intervention: day 0:- Subjects will come fasting for this visit. Urine will be collected. CGM and it's related supplies will be collected back. Records of blood glucose concentrations monitored by finger stick and CGM for the previous 14 days will be obtained to assess their glycemic control while on liraglutide and insulin treatment. They will undergo a meal challenge test (described below). Fructosamine assay will be done on this day. Two questionnaires namely DSQOLS (Diabetes Specific Quality of Life Scale) and PAID (problem areas in Diabetes survey) will be completed. Dapagliflozin or placebo at 5 mg will be started the day after their meal challenge test. Careful adjustments will be made to insulin doses at the discretion of the investigators on the basis of the glucose data obtained from the patients. The target blood glucose will be 70-180 mg/dl at all times of the day and night without increasing the incidence of blood glucose < 70mg/dl. Patients will return to the center after 7 days. Subjects will be asked to make a follow-up appointment with their primary care physician or their endocrinologist a week after the completion of the study i.e. Visit 12(Day 84) to maintain continuity of care and to ensure smooth transition.

Visit 4: Study Intervention day 7:- Insulin dose will be adjusted based on fingerstick blood glucose. Patients will be assessed for any untoward adverse effects with the use of study drug. The dose of dapagliflozin (or placebo) will be increased to 10 mg daily based on investigator's discretion and blood glucose readings.

Visits 5-10: Study Interventions days 14, 21, 35, 49, and 63,70:- Records of blood glucose concentrations of the last 7 days for visit 5 and 6 and for the last 14 days for all other visits will be collected. Insulin dose will be adjusted at the discretion of the study investigator to optimize blood sugar control as per the targets mentioned above on day 0 visit. Any adverse effects with study drug will be assessed. The dose of dapagliflozin (or placebo) will be increased to 10 mg daily based on investigator's discretion if they are still on the starting dose (i.e. 5 mg of dapagliflozin) at the time of visit 5, 6 and 7 only. No further increase in dose of these medications will be made after visit 6. CGM will be fitted on day 70 and will stay on for 2 weeks till day 84.

Visit 11 (Day 77):

CGM will be fitted on this day and will stay on for 2 weeks till day 84. A urine container to collect urine for 24 hours to measure 24-hour urinary glucose will be provided. They will bring the urine specimen with them on Day 84. Subjects will be allowed to conduct this intervention anytime between Day 77 and Day 82 if they choose so.

Visit 12: Study Intervention (day 84). Subjects will come fasting for this visit. Records of blood glucose concentrations monitored by finger stick or CGM for the previous 7 days will be obtained to assess their glycemic control. They will undergo meal challenge test (described below). Two questionnaires namely DSQOLS and PAID will be completed. CGM and related supplies and 24 hour urinary specimen will be collected back. After this visit, subjects will be discharged from the study. Labs will be drawn to measure CBC, comprehensive metabolic panel, Hba1c, Fructosamine and lipid profile. Careful insulin adjustments will be made at the discretion of the investigator depending upon if they choose to continue with liraglutide and or dapagliflozin to optimize blood sugars.

Meal challenge test:- In order to assess the changes induced by dapagliflozin compared to placebo, a meal challenge will be carried before and at the end of the study (day 0 and day 84). (910 Calorie High fat High carbohydrate meal as in several of our previous papers). Dapagliflozin final dose will be administered only on day 84 (45 min prior to the meal). Sequential blood samples will be obtained at 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 and 300 min. Samples at 15, 30, 45, 90, 150 and 210 min will be 5 ml while those at 0, 60, 120, 180, 240 and 300 min will be 30 ml (total volume=210 ml). Blood will be collected from an indwelling intravenous canula in a superficial forearm vein.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus: Fasting c-peptide < 0.1nmol/l on insulin therapy for more than 12 months with or without history of diabetic ketoacidosis and treatment with liraglutide at maximal tolerated doses for at least 6 months prior to start of the study.
* Willing to use a continuous glucose monitoring device (CGM) and regularly measuring their blood sugars four times daily
* HbA1c of less than or equal to 11%.
* Well versed with carbohydrate counting
* Age 18-75 years

Exclusion Criteria:

* Type 1 diabetes for less than 12 months.
* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks
* Hepatic disease (transaminase > 3 times normal) or cirrhosis
* ESRD on hemodialysis; and or e-GFR less than 30 ml/min/1.73m2
* HIV or Hepatitis C positive status
* Participation in any other concurrent clinical trial
* Any other life-threatening, non-cardiac disease
* Use of an investigational agent or therapeutic regimen within 30 days of study
* History of pancreatitis
* Pregnancy
* Inability to give informed consent
* History of gastroparesis
* History of medullary thyroid carcinoma or MEN 2 syndrome
* Family history of MEN 2, Family history of medullary thyroid cancer, or familial medullary thyroid cancer
* Women of childbearing potential who are not using adequate contraception
* Women who are pregnant
* History of serious hypersensitivity reaction to these agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitesh D Kuhadiya, MD, MPH, Principal Investigator — University at Buffalo
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

REFERENCES:
- [Derived] Kuhadiya ND, Ghanim H, Mehta A, Garg M, Khan S, Hejna J, Torre B, Makdissi A, Chaudhuri A, Batra M, Dandona P. Dapagliflozin as Additional Treatment to Liraglutide and Insulin in Patients With Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Sep;101(9):3506-15. doi: 10.1210/jc.2016-1451. Epub 2016 Aug 4. PMID 27490915

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 12 weeks of treatment with Insulin, Liraglutide and "Dapagliflozin Placebo"
  Insulin
  Liraglutide: Victoza(Liraglutide) is a GLP-1 agent.
  Dapagliflozin placebo: Dapagliflozin placebo looking similar to active drug Dapagliflozin in external appearance but not containing active ingredient dapagliflozin
- Active Drugs: 12 weeks of treatment with Insulin, Liraglutide and "Active Dapagliflozin Drug"
  Dapagliflozin: Dapagliflozin or Farxiga is a SGLT-2 inhibitor
  Insulin
  Liraglutide: Victoza(Liraglutide) is a GLP-1 agent.
Period: Overall Study
Arm/Group | Placebo | Active Drugs
Started | 9 | 17
Completed | 9 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drugs | Total
Number analyzed (Participants) | 9 | 17 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (3) | 55 (3) | 53 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 3 | 7 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HbA1c % [Mean (Standard Deviation); unit: %] | 7.4 (0.2) | 7.8 (0.2) | 7.6 (0.2)
Average glucose [Mean (Standard Deviation); unit: mmol/L] | 9.32 (0.49) | 9.16 (0.38) | 9.24 (0.41)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change After 12 Weeks From Baseline in Mean HbA1c With Addition of Dapagliflozin Compared to Placebo.
Description: T1D. Conservatively estimating a difference in mean HbA1c (the primary end point) of 0.5% before and after the treatment, and a sample size of 30 (2:1 drug to placebo ratio) should provide adequate power (.8) to detect a significant difference (.05) provided the standard deviation of the residuals in not greater than 0.4%. The sample size includes an additional 20% to account for the potential dropout.
  Changes in these end points were calculated by averaging the differences in weekly average values from baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: % HbA1c
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
% HbA1c | 0 (0.2) | -0.66 (0.1)

2. Secondary Outcome: Change in Time Spent at Normal Glucose Concentrations Between 70-160mg/dl
Description: Comparison of the change in time spent at normal glucose concentrations between 70-180mg/dl after treatment with 12 weeks of dapagliflozin in addition to liraglutide and insulin.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
percentage of time | -1.4 (1.0) | 10 (4)

3. Secondary Outcome: Change in 24-hour Urine Glucose Excretion.
Description: Comparison of change in 24-hour urine glucose excretion after 12 weeks of treatment of dapagliflozin in addition to liraglutide and insulin compared to baseline.
Time Frame: 12 weeks.
Measure: Mean (Standard Error); unit: gram/day
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
gram/day | 2.1 (1.1) | 66.9 (4.7)

4. Secondary Outcome: Change in Total Daily Insulin Requirements
Description: Comparison of the change from baseline in total daily insulin requirements in units per kilogram after treatment 12 weeks of dapagliflozin or placebo in addition to liraglutide and insulin.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Units/Kg
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
Units/Kg | -0.1 (2.4) | -3.5 (1.9)

5. Secondary Outcome: Change in Body Weight
Description: Comparison of change from baseline in Body weight after 12 weeks treatment with dapagliflozin or placebo in addition to liraglutide and insulin.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
Kg | 0.7 (1.5) | -1.9 (0.5)

6. Secondary Outcome: Change in Systolic Blood Pressure Before and After Treatment
Description: Comparison of Systolic blood pressure in mm Hg before and after 12 weeks treatment with dapagliflozin in addition to liraglutide and insulin.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
mmHg | -2 (3) | -12 (4)

7. Secondary Outcome: Change in Blood Ketone Bodies
Description: change from baseline in blood ketone bodies (measured as beta-hydroxybutyrates) after 12 weeks treatment with dapagliflozin or placebo in addition to liraglutide and insulin.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mM
Arm/Group | Placebo | Active Drugs
Number analyzed (Participants) | 9 | 17
mM | -0.03 (0.06) | 0.20 (0.09)

ADVERSE EVENTS:
Time Frame: 12 WEEKS
Arm/Group | Placebo | Active Drugs
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/17
Other Adverse Events (participants affected / at risk) | 0/9 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Active Drugs (N=17)
DKA (Endocrine disorders) | 0 | 2 (2) — Two patients suffered from diabetic ketoacidosis within a day after increasing the dose of dapagliflozin to 10mg and were withdrawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes